CLINICAL TRIAL: NCT04334122
Title: The Efficacy Of Instrument-Assisted Soft Tissue Mobilization At Lumbar Region Disc Herniations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Ali Yıldırım, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bvuayildirim
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Lumbar Disc Herniation; Instrument-assisted Soft Tissue Mobilization
Keywords: pain; instrument-assisted soft tissue mobilization; depression; functionality; lumbar disc herniation; quality of life
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): All patients in the control group were given a traditional physiotherapy program applied in lumbar disc herniation for 4 weeks (20 sessions) and 5 days a week.
  As a traditional treatment, patients received hot packs, conventional transcutaneous electrical nerve stimulation (TENS), therapeutic ultrasound and exercise.
  Hot packs used as superficial heat were wrapped in a towel and applied to the waist area for 20 minutes.
  Conventional TENS used as analgesic current were applied to the waist region for 20 minutes with 4 electrodes with 2 outputs, with a current time of 180 ms at a frequency of 80 Hz.
  It was applied with a dose of 1Mhz for 5 minutes with ultrasan (Chattanooga Intelect Mobile Combo model device) used to heat deep tissues.
  Waist exercises were asked to be done during the treatment, with 10 repetitions, each exercise twice a day (morning and evening).
  Interventions: Other: Traditional physiotherapy
- Experiment group (Experimental): In addition to the traditional physiotherapy program, tool-assisted soft tissue mobilization was performed 3 times a week (12 sessions with 1 day interval) in the experimental group.
  Instrument Assisted Soft Tissue Mobilization (IASTM) treatment was applied to ilicostalis lumborum, priformism, gluteus medius, erector spinas, quadratus lumborum muscles, superficial and deep fascia. Before applying the application, petroleum jelly was applied to the area and the tool was slipped.
  IASTM treatment was applied to the treated muscle fibers for 6 minutes, each technique (SWEEP-FAN-BRUSH-SWEEP techniques) with 8-10 repetitions.
  Sweep: Applied in all directions at 30 or 60 degree angle. Fan: It was applied by moving one side fixed arm at 30 degree angle. Brush: It was applied in straight steps at 30 degrees angle. Each stage of IASTM treatment was done by the physiotherapist.
  Interventions: Other: Instrument-assisted soft tisue mobilization; Other: Traditional physiotherapy

INTERVENTIONS:
Other: Instrument-assisted soft tisue mobilization — All patients in the experimental group were given a traditional physiotherapy program applied in lumbar disc herniation for 4 weeks (20 sessions) and 5 days a week.
  In addition to the traditional physiotherapy program, the patients in the experimental group were subjected to tool-assisted soft tissue mobilization 3 times a week (12 sessions with 1 day interval).
  All evaluations were repeated to all patients in the experimental and control groups after four weeks.
  Arms: Experiment group
Other: Traditional physiotherapy — All patients in the control group were given a traditional physiotherapy program applied in lumbar disc herniation for 4 weeks (20 sessions) and 5 days a week.

SUMMARY:
This study was carried out to investigate the effect of instrument-assisted soft tissue mobilization in patients with lomber region disc herniation. 60 patients with lumbar disc herniation between the ages of 30-65 were included in the study. Following the evaluation, the patients were divided into two groups by closed envelope method; control group (n=30) and experimental group (n=30). In both groups, 4 weeks (20 sessions) hot pack (hotpack), conventional transcutaneous electrical nerve stimulation (TENS), therapeutic physical therapy program with therapeutic ultrasound applications were performed. In addition to this program, Instrumental Assisted Soft Tissue Mobilization (IASTM) was applied to the experimental group in 12 sessions of 3 times a week. This technique was performed by using stainless steel tools of different sizes and shapes. IASTM treatment was performed (including SWEEP-FAN-BRUSH-SWEEP technique, 45° angle with the skin, by 8-10 repetitions) for the ilicostalis lumborum, priformis, gluteus medius, erector spines, quadratus lumborum muscles, superficial and deep fascia. Depression levels of the patients were evaluated with Beck Depression Scale, before the treatment and after 4 weeks pain severity, VAS pain scale, functional status with Oswestry Scale, quality of life with Short Form-36 (SF-

36) and normal range of motion with goniometer. The results were analyzed by using SPSS v.20 program. In all analyzes, the significance ratio was accepted as p <0.05. At the end of the four-week treatment program, significant improvements were observed in VAS levels, normal joint movements (flexion, extension, right-left lateral flexion, rotation) in both groups (p <0.05). Oswestry and Beck Depression Scale scores showed significant improvement merely in the experimental group compared to the control group (p <0.05). There was no significant difference in VAS values, normal joint motion and Oswestry scale while there was no notable difference in SF-36 and Beck Depression Scale. As a result of the study, it was concluded that IASTM is a more effective method on normal range of motion and functionality in comparison with traditional physiotherapy program in patients with lumbar disc herniation and it can be used as an alternative method in patients during the physiotherapy and rehabilitation program if needed.

ELIGIBILITY:
Inclusion Criteria:

1. Bulging and protruding disc presence
2. Facet joint problem
3. Mechanical low back pain

Exclusion Criteria:

1. Extruded and sequestrated disc presence
2. Previous operational status through the lumbar region
3. Having inflammatory pain (osteoarthritis)
4. Pain associated with malignancy (primary or metastatic tumors)
5. Severe psychological discomfort
6. Having communication problems

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Demographic information | 4 week
  Personal information (name, surname, address, telephone, marital status, educational status, occupational and health security), demographic and clinical information (age (year), gender, height (cm), weight (kg), BMI of all patients participating in the study (calculated by the formula of the ratio of body weight to neck squared (kg / m²)), information about the disease, drugs used for lumbar disc hernia, other drugs used, presence of chronic disease, surgical history, smoking and alcohol use] by questioning '' Demographic Information Forms '' recorded.
Assessment of pain (VAS) | 4 week
  The pain intensities of the patients at rest, during the activity and at night were determined using the Visual Analogue Scale (VAS). VAS is an easy-to-apply scale, as values that cannot be measured numerically can be digitized and quickly understood.
  The patients were asked to mark their severity (rest, activity, night) on a 10 cm line. The starting point of the truth was '' 0 '' '' I have no pain '', the end point was '' 10 '' '' I have pain of unbearable severity ''. The point that the patient marked on the right was measured with a ruler and recorded in "cm". Localization of the pain, its frequency and the causes that increase and decrease pain were questioned and recorded. The Turkish validity and reliability study of the scale was performed.
Evaluation of normal joint motion (NEH) | 4 week
  The limitation of flexion, extension, lateral flexion and rotation movements of the lumbosacral joint was measured using a universal goniometer. All normal joint movements were repeated 3 times and the average of the obtained values was recorded in degrees.
Evaluation of the quality of life | 4 week
  Quality of life was assessed with the survey "SF-36 (Short form-36) quality of life". SF-36 is a generic scale that evaluates the overall health status. It consists of 36 questions that evaluate 2 main (physical and mental component) and 8 sub parameters (physical function, emotional function, physical role, social function, mental health, pain, general health and vitality). The score of each subgroup is evaluated between 0-100. A high score indicates that the quality of life is good. The Turkish validity and reliability study of the SF-36 questionnaire was conducted.
Evaluation of depression | 4 week
  Depression level of the patients was evaluated by Beck Depression questionnaire. The scale developed by Beck consists of 21 questions. 4-point Likert scoring is used in the scale. Each item gets points between 0-3. The total score ranges from 0-63.
  Points obtained from the survey;
  0-10 points → no depression
  11-17 points → mild depression
  18-23 points → moderate depression
  24 points above → interpreted as severe depression.
  The Turkish validity and reliability study of the scale was conducted.
Functional evaluation for low back pain | 4 week
  Oswestry Disability Index was used to evaluate the disability caused by low back pain. The scale evaluates how much back pain affects daily life activities. Pain severity consists of 10 questions evaluating personal care, weight lifting, walking, sitting, standing, sleep quality, social life, ability to travel and the degree of pain. Six-point likert scoring is used. A high total score indicates an increase in disability. The Turkish validity and reliability study of this scale was conducted.
  Points obtained from the survey;
  0% - 20% → minimal disability
  20% to 40% → mild disability
  40% to 60% → severe disability
  60% - 80% → complete limitation
  80% - 100% → bed-dependent (or symptoms are exaggerated)

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided